CLINICAL TRIAL: NCT02381015
Title: Clinical Validity and Utility of Genomic-targeted Chemoprevention of PCa: Aim 4a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Van Andel Research Institute (Other); Spectrum Health Medical Group (Unknown); National Cancer Institute (NCI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Jianfeng Xu, Professor of Human Genomics and Personalized Medicine, Epidemiology, Cancer Biology, and Urology, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00011784; 1RC2CA148463-01 (NIH)
Record Dates: First submitted 2015-02-28; First posted 2015-03-06 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer; Prostate Cancer, Familial; Hereditary Prostate Cancer
Keywords: Genetic testing; Genomic testing; Chemoprevention; Prostate Specific Antigen; Prostate Cancer; Predictive Genetic Testing; Genetic Counseling; Prostate-Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms; Prostate cancer, familial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Genetic Risk Score: Number Format (Experimental): Genetic Risk Score: Number Format Subjects receive genetic risk scores in a number format.
  Interventions: Genetic: Genetic Risk Score: Number Format
- Genetic Risk Score: Number + Pictograph (Experimental): Genetic Risk Score: Number + Pictograph Subjects receive genetic risk scores in a number and pictograph format.
  Interventions: Genetic: Genetic Risk Score: Number + Pictograph
- Family History: Number Format (Experimental): Family History: Number Format Subjects receive family history risk in a number format.
  Interventions: Behavioral: Family History: Number Format
- Family History: Number + Pictograph (Experimental): Family History: Number + Pictograph Subjects receive family history risk in a number and pictograph format.
  Interventions: Behavioral: Family History: Number + Pictograph

INTERVENTIONS:
Genetic: Genetic Risk Score: Number Format — Genetic Risk Score: Number + Pictograph Genetic risk score based on validated panel of 46 single nucleotide polymorphisms previously identified to be associated with Prostate Cancer risk by Genome Wide Association Studies, presented to subjects as a number.
  Arms: Genetic Risk Score: Number Format
Genetic: Genetic Risk Score: Number + Pictograph — Genetic Risk Score: Number + Pictograph Risk information conveyed as either a number or a number + pictograph, depending on randomization group.
  Arms: Genetic Risk Score: Number + Pictograph
Behavioral: Family History: Number Format — Family History: Number Format Risk information conveyed as either a number or a number + pictograph, depending on randomization group.
  Arms: Family History: Number Format
Behavioral: Family History: Number + Pictograph — Family History: Number + Pictograph Risk information conveyed as either a number or a number + pictograph, depending on randomization group.
  Arms: Family History: Number + Pictograph

SUMMARY:
This study was designed to compare the efficacy, perception, decision making, and cost-effectiveness of genomic and non-genomic approaches for risk assessment of prostate cancer and for chemoprevention of prostate cancer.

DETAILED DESCRIPTION:
ABSTRACT: This clinical trial registration is focused on Aim 4 within the overall project described in the following.

Prostate cancer (PCa) is the most common cancer among men in the U.S. One important strategy to address this public health concern is to prevent the disease. Two large randomized clinical trials, The Prostate Cancer Prevention Trial (PCPT) and The Reduction by Dutasteride of Prostate Cancer Events (REDUCE), have demonstrated a 23-25% reduction in PCa risk with the use of 5 alpha reductase inhibitors (5ARIs: finasteride and dutasteride). However, 5ARIs have not been widely adopted due, in part, to poor cost-effectiveness. We hypothesize that targeted chemoprevention, based on 1) overall genetic risk [family history (FH) and PCa risk-associated genetic variants], and 2) polymorphisms that interact with 5ARIs, may be more efficacious and cost-effective, and thus more likely to be employed by physicians and their patients. The effectiveness of this genomic-targeted approach needs to be systematically evaluated and compared to non-genomic approaches using evidence-based methods such as those recommended by the EGAPP (Evaluation of Genomic Applications in Practice and Prevention) working group. We have assembled a multidisciplinary research team to address an overarching question of whether a genomic-targeted approach improves outcomes related to chemoprevention of PCa using 5ARIs compared to a non-targeted approach. We will evaluate and compare the efficacy, perception, decision making, and cost-effectiveness of genomic and non-genomic approaches in two existing large randomized clinical trials (Reduction by Dutasteride of Prostate Cancer Events (REDUCE) and Prostate Cancer Prevention Trial (PCPT)), two new study populations of men at risk for PCa, and in a survey of physicians. The unique study design of REDUCE and PCPT, with end-of-study prostate biopsies, allows us to address two critical questions in this study: Prostate Specific Antigen (PSA) detection-bias of PCa risk-associated Single Nucleotide Polymorphisms (SNPs) and efficacy of genomic-targeted chemoprevention of PCa using 5ARIs. We have the following specific aims: 1) assess the clinical validity of PCa risk prediction models using a panel of non PSA detection biased PCa risk-associated SNPs. 2) identify and assess the clinical validity of novel polymorphisms that interact with 5ARIs in reducing PCa diagnosis using both genome-wide and candidate gene approaches, 3) assess the clinical utility of a genomic-targeted approach by comparing its reduction in rates of PCa with non-targeted chemoprevention, 4) compare perception and decision making of physicians and patients for genomic and non-genomic-targeted chemoprevention of PCa, and 5) Compare the cost-effectiveness of genomic and non-genomic-targeted chemoprevention of PCa. Results from this study will provide comprehensive data for evidence-based evaluation by the Center for Disease Control's Evaluation of Genomic Applications in Practice and Prevention (EGAPP) working group, provide a proof of principle study of Comparative Effectiveness Research (CER), and will help build a road map for future Genomic and Personalized Medicine (GPM) in the 21st century.

ELIGIBILITY:
Inclusion Criteria:

* age 40 to 49 years, self-defined Caucasian background, and no prior prostate specific antigen (PSA) screening nor prostate cancer (PCa) diagnosis.

Exclusion Criteria:

* outside of age range, or not self defined Caucasian background, or a prior history of PSA screening or PCa diagnosis

Ages: 40 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xu, Dr.P.H., Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
There is no intent to share individual participant data (IPD). The terms included in the study consent form do not allow sharing of IPD.

RESULTS

PARTICIPANT FLOW:
Period: Visit 1 - Enrollment
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Started | 175 | 175 | 175 | 175
Completed | 175 | 173 | 175 | 172
Not Completed | 0 | 2 | 0 | 3
Period: Visit 2 - Results DIsclosure
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Started | 175 | 173 | 175 | 172
Completed | 172 | 168 | 173 | 169
Not Completed | 3 | 5 | 2 | 3
Period: Visit 3 - 3 Months Followup
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Started | 172 | 168 | 173 | 169
Completed | 172 | 168 | 173 | 169
Not Completed | 0 | 0 | 0 | 0
Period: Year 3 Chart Review
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Started | 172 | 168 | 173 | 169
Completed | 125 | 134 | 115 | 118
Not Completed | 47 | 34 | 58 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph | Total
Number analyzed (Participants) | 175 | 175 | 175 | 175 | 700
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (2.85) | 44.8 (3.06) | 44.7 (2.84) | 45.0 (2.76) | 44.85 (2.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 175 | 175 | 175 | 175 | 700
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 175 | 175 | 175 | 175 | 700
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — United States, Western Michigan
  participants
    United States | 175 | 175 | 175 | 175 | 700

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Prostate Specific Antigen (PSA) Discussion With Physician at 3 Months, Measured by Survey
Description: Discussion with Physician regarding PSA screening, measured by survey 3 months after provision of risk information
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 175 | 173 | 175 | 172
participants | 34 | 30 | 25 | 22
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; Test type: Superiority or Other; p = 0.29, Chi-squared

2. Primary Outcome: Number of Participants Who Had PSA Testing at 3 Months, Measured by Survey
Description: PSA screening, measured by survey 3 months after provision of risk information.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 172 | 168 | 173 | 169
participants | 8 | 7 | 4 | 3
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; Test type: Superiority or Other; p = 0.35, Chi-squared

3. Primary Outcome: Number of Participants Who Had PSA Testing at 3 Years, Measured by Medical Records
Description: PSA screening, measured by medical records 3 years after provision of risk information.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 125 | 134 | 115 | 118
participants | 45 | 46 | 29 | 40
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; Test type: Superiority or Other; p = 0.29, Chi-squared

4. Secondary Outcome: Anxiety, Measured by State-trait Anxiety Inventory (STAI)
Description: Immediate reaction to risk information. Measured by state anxiety scale that assess current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. A shortened version of questions 1,3,5,9,11,12,13,15,17, and 19 from STAI form XI were used. Each item, within then STAI is scored on a scale of 1-4 and with 10 items, the possible range of total scores was 10 (lowest anxiety) to 40 (highest anxiety). Lowest scores represent better outcomes.
Time Frame: Baseline
Population: Computerized randomization of 700 study identifiers into 175 blocks of four each was completed prior to enrollment. Genetic Risk Score=GRS and Family History=FH. Randomization groups were (Group 1) GRS+FH as a number; (Group 2) GRS+FH as a number and pictograph; (Group 3) FH as a number; and (Group 4) FH as a number and pictograph.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 175 | 172 | 174 | 171
units on a scale | 15.25 (4.43) | 15.95 (5.19) | 14.92 (4.40) | 15.12 (3.93)
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; Test type: Superiority or Other; p = 0.49, Kruskal-Wallis

5. Secondary Outcome: Accuracy of Immediate Recall of Risk Information Measured by Survey
Description: Mean between Immediate recall of risk information and told risk information. Immediate recall is measured by survey question: "Based on the information given to you, what were you told is your chance of developing prostate cancer in your lifetime from 0% to 100% ______ %"
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage of recall
Groups:
- Genetic Risk Score: Number Format: Genetic Risk Score: Number Format Subjects receive genetic risk scores in a number format. Genetic risk score based on validated panel of 46 single nucleotide polymorphisms previously identified to be associated with Prostate Cancer risk by Genome Wide Association Studies, presented to subjects as a number. Data presented as linear relationship between told risk and immediate recall.
- Genetic Risk Score: Number + Pictograph: Genetic Risk Score: Number + Pictograph Subjects receive genetic risk scores in a number and pictograph format. Genetic Risk Score: Number + Pictograph: Genetic Risk Score: Number + Pictograph Risk information conveyed as either a number or a number + pictograph, depending on randomization group. Data presented as linear relationship between told risk and immediated recall.
- Family History: Number Format: Family History: Number Format Subjects receive family history risk in a number format. Family History: Number Format: Family History: Number Format Risk information conveyed as either a number or a number + pictograph, depending on randomization group. Data presented as linear relationship between told risk and immediated recall.
- Family History: Number + Pictograph: Family History: Number + Pictograph Subjects receive family history risk in a number and pictograph format. Family History: Number + Pictograph: Family History: Number + Pictograph Risk information conveyed as either a number or a number + pictograph, depending on randomization group. Data presented as linear relationship between told risk and immediated recall.
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 175 | 173 | 174 | 173
Percentage of recall | 0.65 (4.05) | 0.72 (3.84) | 0.26 (1.42) | 1.0 (5.84)
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; The statistical analysis shows the relation between risk given and risk recall at the immediate post results assessment for the total number of participants; Test type: Other; p = 0.42, ANOVA; Beta = 93.5, Standard Error of Mean 1.55

6. Secondary Outcome: Accuracy of Recall of Risk Information at 3 Months Measured by Survey
Description: Mean between recall of risk information at 3 months measured by survey, and told risk information. Recall at 3 months is measured by survey question: "Based on the information given to you, what were you told is your chance of developing prostate cancer in your lifetime from 0% to 100% ______ %"
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: Percentage of recall
Groups:
- Genetic Risk Score: Number Format: Genetic Risk Score: Number Format Subjects receive genetic risk scores in a number format. Genetic risk score based on validated panel of 46 single nucleotide polymorphisms previously identified to be associated with Prostate Cancer risk by Genome Wide Association Studies, presented to subjects as a number. Data presented as linear relationship between told risk and immediated recall.
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Number analyzed (Participants) | 172 | 168 | 173 | 169
Percentage of recall | 3.30 (6.04) | 3.78 (6.01) | 4.43 (6.92) | 4.38 (7.33)
Statistical Analysis 1: Comparison: Genetic Risk Score: Number Format vs Genetic Risk Score: Number + Pictograph vs Family History: Number Format vs Family History: Number + Pictograph; Test type: Other; p = 0.33, ANOVA; Beta = 94.7, Standard Error of Mean 2.93

ADVERSE EVENTS:
Arm/Group | Genetic Risk Score: Number Format | Genetic Risk Score: Number + Pictograph | Family History: Number Format | Family History: Number + Pictograph
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175 | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175 | 0/175 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No